CLINICAL TRIAL: NCT02466451
Title: Observational Longitudinal Study in Children With the Diagnosis of Diaphragmatic Hernia and/or Oesophageal Atresia for Assessing Lung Function Parameters and Quality of Life
Brief Title: Study in Children With the Diagnosis of Congenital Diaphragmatic Hernia (CDH) and Oesophageal Atresia (EA)
Acronym: CDH-EA
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Senior Researcher, Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 5/2012
Record Dates: First submitted 2015-05-12; First posted 2015-06-09 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Diaphragmatic Hernia; Oesophageal Atresia
MeSH Terms: conditions — Hernia, Diaphragmatic; Esophageal Atresia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children operated at birth on CDH and EA: Standardized Questionnaires:For not collaborative patients,< 4 years:Standardized questionnaire collecting anamnestic-clinical data;Stress Parenting Index questionnaire and COPE brief questionnaire(Questionnaire assessing adaptation strategies of parents) For collaborative patients, >4 years:Standardized questionnaire collecting anamnestic-clinical data;Fractional exhaled nitric oxide (FeNO) assessment (oral and alveolar);Spirometry;6-minutes walk test (WT 6'); Prick tests;Children Quality of life questionnaire (KINDL questionnaire);Psychological test (Raven Matrices);Stress Parenting Index questionnaire and COPE brief questionnaire (Questionnaire assessing adaptation strategies of parents).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — For not collaborative patients, under the age of 4 years:
  * Standardized questionnaire collecting anamnestic-clinical data
  * Stress Parenting Index questionnaire and COPE brief questionnaire(Questionnaire assessing adaptation strategies of parents).
  For collaborative patients, over the age of 4 years:
  * Standardized questionnaire collecting anamnestic-clinical data
  * Fractional exhaled nitric oxide (FeNO) assessment (oral and alveolar )
  * Spirometry
  * 6-minutes walk test (WT 6')
  * Prick tests
  * Children Quality of life questionnaire (KINDL questionnaire)
  * Psychological test (Raven Matrices)
  * Stress Parenting Index questionnaire and COPE brief questionnaire (Questionnaire assessing adaptation strategies of parents)
  Other Names: Standardized Questionnaires

SUMMARY:
Observational longitudinal study in children operated at birth on diaphragmatic hernia and/or oesophageal atresia : assessment of lung function parameters; assessment of quality of life and cognitive development; assessment of stress parenting and strategies of adaptation.

DETAILED DESCRIPTION:
Observational longitudinal study in children operated at birth on diaphragmatic hernia and/or oesophageal atresia : assessment of lung function parameters; assessment of quality of life and cognitive development; assessment of stress parenting and strategies of adaptation.

Tools: Anamnestic-clinical questionnaire, Spirometry, Plethysmography, Fractional exhaled nitric oxide (FeNO) assessment (oral and alveolar ), 6-minutes walk test (WT 6'), Prick tests, Quality of life in children questionnaire(KINDL, quality of life), Psychological test for cognitive development (Raven Matrices)

ELIGIBILITY:
Inclusion Criteria:

* Children operated at birth on diaphragmatic hernia and/or oesophageal atresia
* Written informed consent, signed by parents

Exclusion Criteria:

* Children that have had infections in the last 4 weeks
* Children with ongoing diseases
* Children that take drugs able to modify the lung function

Ages: 5 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 33 Children operated at birth on diaphragmatic hernia and/or oesophageal atresia (age range : 5 months - 12 years old)
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | 1 year
  Spirometry

SECONDARY OUTCOMES:
Quality of Life | 1 year
  QoL Questionnaire